CLINICAL TRIAL: NCT02531269
Title: Effectiveness Of Daclatasvir-Based Regimens In Patients With Chronic Hepatitis C Infection In Europe: Experience From Named Patient Program And From Early Post-Marketing Authorization Period
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Basel Institute of Clinical Epidemiology (BICE) (Other)
Responsible Party: Sponsor
Other Study IDs: AI444-319
Record Dates: First submitted 2015-08-11; First posted 2015-08-24 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients treated with DCV (NPP)+Sofosbuvir +/- Ribavirin (RBV)
- Patients treated with DCV (NPP) + Simeprevir +/- RBV
- Patients treated with DCV(post-marketing) + Sofosbuvir +/- RBV
- Patients treated with DCV(post-marketing) + Simeprevir +/- RBV

SUMMARY:
Using European data from patients included in the Named Patient Program (NPP) and from the early post-marketing authorization period, the present study aims to describe patient characteristics and to describe the effectiveness of Daclatasvir (DCV)-based regimens in Europe. This will be a retrospective cohort study of patients who received treatment with a DCV-based regimen in the following context:

* Patients enrolled within the European NPP in one of the following countries Austria, Denmark, Italy, Sweden, Spain, Switzerland, United Kingdom; or
* In those countries where DCV is commercially available (ie, Sweden, Germany, United Kingdom), patients who received DCV during the early post-marketing authorization period

The results of this study will contribute to a better understanding of effectiveness of DCV-based regimens in a population that differs from population in the clinical trials, and therefore will provide additional valuable information to inform clinical practice.

This study intends to estimate primarily the effectiveness of DCV-based regimens as measured by the sustained virologic response at post treatment follow-up visit week 12 (SVR12). As well as estimate the effectiveness of DCV-based regimens as measured by SVR12 after the end of Hepatitis C virus (HCV).

This study intends also to describe as secondary objectives the characteristics (ie, demographic and clinical characteristics and treatment patterns of patients starting a new DCV-based regimens) of patients receiving DCV as well as the effectiveness of DCV-based regimens as measured by:

* On-treatment virological response at post treatment follow-up visit Week 4; and
* Virological response at the end of treatment (EOT); and
* The sustained viral response at post treatment follow-up visit Week 4 (SVR4) and post treatment follow-up visit Week 24 (SVR24); and
* The occurrence of virological failure (on-treatment and relapse).

An exploratory objective will be to assess the concordance between SVR4 and SVR12 among the overall population treated with DCV.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in the DCV NPP from 7 European countries (Austria, Denmark, Italy, Sweden, Spain, Switzerland, and UK). The following patients were eligible to participate in the NPP

  * The patient have a serious or life-threatening condition that is impacting life expectancy within 12 months.
  * There are no comparable or satisfactory alternative treatments options exist for the patient, and/or currently available treatment options have been exhausted.
  * The patient was ineligible to participate in a clinical trial, or there was no ongoing clinical trial in the patient´s country of residence to treat his/her HCV-infection.
* In countries where DCV is commercially available at time of study initiation(Sweden, UK, and Germany), patients treated with DCV during the early post-marketing authorization period.
* Patients initiating any DCV-based regimen during the inclusion periods.
* Recorded in one of the HCV data sources used for the study.

Exclusion Criteria:

* Patients included in the DCV Compassionate use program (CUP) (AI444-237 Protocol) open in 6 European countries (Germany, Austria, Sweden, Netherlands, Norway and UK) after Committee for Medicinal Products for Human Use (CHMP) opinion for the DCV CUP in Europe will be excluded since these patients will be analyzed as part of separate datasets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from European HCV registries or databases in specific health-care facilities from Austria, Denmark, Italy, Sweden, Spain, Switzerland, and United Kingdom (UK)
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
SVR12 | Up to 36 months
  Effectiveness of DCV-based regimens as measured by the SVR12, overall and in specific patient sub-populations

SECONDARY OUTCOMES:
SVR4 | Up to 36 months
  Effectiveness of DCV-based regimens as measured by SVR4
SVR24 | Up to 36 months
  Effectiveness of DCV-based regimens as measured by SVR24
On-treatment Virological response at week 4 assessed by measuring viral load | Up to 36 months
Virological response at the end of treatment (EOT) assessed by measuring viral load | Up to 36 months
The occurrence of virological failure (on-treatment and relapse) assessed by measuring viral load | Up to 36 months
  Virological failure is defined as virologic breakthrough, other on-treatment failure or relapse, where:
  * Virologic breakthrough is defined as confirmed ≥ 1 log10 IU/mL HCV RNA on treatment increase from nadir, or confirmed increase in HCV RNA ≥ LLOQ if HCV RNA previously declined to < LLOQ (TD/TND). (LLOQ: Lower limit of quantification)
  * Relapse is defined as HCV RNA < LLOQ (TND) at End of Treatment followed by confirmed detectable HCV RNA ≥ LLOQ in any follow-up visit window.
  * On-treatment failure is defined as HCV RNA ≥ LLOQ at any time point not meeting the definition of virologic breakthrough or relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Basel, Switzerland

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx